CLINICAL TRIAL: NCT06613425
Title: Combined Platelet Transfusion:A Single-arm, Open, Prospective, Non-inferiority Clinical Trial
Brief Title: Clinical Study of Combined Platelet Transfusion
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The General Hospital of Western Theater Command (Other)
Responsible Party: Principal Investigator, zhang li, PHD，Professor, The General Hospital of Western Theater Command
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024EC4-ky004
Record Dates: First submitted 2024-08-28; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Hematologic Diseases
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Combined platelet
  Interventions: Combination Product: Combined platelets

INTERVENTIONS:
Combination Product: Combined platelets — 1 therapeutic dose combined platelet contained no less than 2.5 ×10^11 platelets as a quality standard.

SUMMARY:
Platelet transfusion is an irreplaceable and important treatment method for clinical prevention and treatment of thrombocytopenia or platelet dysfunction. Due to various factors, it is difficult to achieve platelet ABO complete homotypic transfusion in clinical practice. When ABO-compatible platelets cannot be obtained, plasma-reduced platelets, platelets with low anti-A or anti-B titers are often used in clinical practice to reduce the risk of ABO-incompatible platelet-compatible transfusion reactions. The combined platelets prepared in this study can achieve ABO primary and secondary side compatible infusion.

DETAILED DESCRIPTION:
Combined platelet transfusion is a single-arm, open, prospective, non-inferiority study initiated by researchers. Patients with hematological diseases who were admitted to the research unit and applied for platelet transfusion within two years were included in the study after informed consent. When the subjects applied for platelet transfusion during the study period, ABO homotype platelet transfusion was preferred. When there was no ABO homotype platelet in the inventory, ABO primary and secondary side compatible combined platelet transfusion was given. The study period was 2 years, including 15 months of enrollment, 6 months of treatment, and 3 months of follow-up after the end of the treatment period

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 18-65 years; 2. Disease treatment in the research hospital; 3. Applied for platelet transfusion therapy.

Exclusion Criteria:

* 1. One month before the start of this study, he participated in other clinical trials of drugs and instruments related to platelet transfusion efficacy; 2. Without platelet transfusion indications; 3. Only received platelet transfusion in the outpatient department and left the hospital without efficacy evaluation after transfusion; 4. Gave up platelet transfusion therapy for any reason after enrollment; 5. Transferred or discharged from hospital for any reason before platelet transfusion after enrollment; 6. Did not receive combined platelet transfusion during the 6-month treatment period after enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-07-29 (Estimated); Study Completion 2025-10-28 (Estimated)

PRIMARY OUTCOMES:
Efficacy evaluation of combined platelet transfusion | From the start of infusion of combined platelets to 6 months later
  The platelet count was measured before blood transfusion and 1 hour and 24 hours after blood transfusion, and the WHO bleeding grade was recorded. The platelet incremental correction index ( CCI ) was calculated at 1 hour and 24 hours after infusion. CCI > 7.5 at 1 hour, CCI > 4.5 at 24 hours, or the control or improvement of WHO bleeding symptoms after infusion were effective for infusion.
  CCI = ( PLT after infusion-PLT before infusion ) × body surface area ( m2 ) × 1000 / total platelet count ( × 1011 ), body surface area = 0.0061 × height ( cm ) + 0.0128 × weight ( Kg ) - 0.1529.
  PPR ( % ) = ( PLT after infusion-PLT before infusion ) × blood volume ( L ) × 100 % / total platelet count × 2 / 3, blood volume = 0.07 × body weight ( Kg ).

SECONDARY OUTCOMES:
Adverse reactions of blood transfusion | From the start of infusion of combined platelets to 6 months later
  During and after blood transfusion, the occurrence time, type, treatment and recovery time of adverse reactions of blood transfusion were collected and recorded, as well as the occurrence time, type, treatment and recovery time of adverse events of blood transfusion.
Safety evaluation of combined platelet transfusion | From the start of infusion of combined platelets to 6 months later
  Blood transfusion-related infectious markers ( HBsAg, HBV DNA, anti-HCV, HCV RNA, HIV Ag / Ab, HIV RNA, anti-TP ) were detected before and after the last blood transfusion.
Platelet antibody screening | From the start of infusion of combined platelets to 6 months later
  Platelet antibodies of the subjects were screened before blood transfusion and at the end of the intermediate follow-up period during infusion.
Adverse events of blood transfusion | From the start of infusion of combined platelets to 6 months later
  The occurrence of adverse transfusion events in the whole process of combined platelet transfusion : time, place, type, measures and consequences.
Waiting time for platelet transfusion | From the start of infusion of combined platelets to 6 months later
  The time from the clinical submission of platelet transfusion application to the start of platelet transfusion
Interval time, frequency and total amount of platelet transfusion | From the start of infusion of combined platelets to 6 months later
  The interval time, frequency and total amount of platelet transfusion in the enrolled group were recorded.
Bleeding adverse events during hospitalization | From the start of infusion of combined platelets to 6 months later
  The number of bleeding, symptoms and treatment measures during hospitalization were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: zhang li, Principal Investigator — The General Hospital of Weastern Theater Command
Locations (1):
- Li Zhang, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No